CLINICAL TRIAL: NCT00752765
Title: The Effects of Bariatric Surgery Weight Loss on Knee Pain in Patients With Osteoarthritis of the Knee
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kevin P. Black, Professor and Chair, Orthopaedics and Rehabilitation, Penn State University
Other Study IDs: 28727
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2012-05

CONDITIONS: Knee Pain; Knee Osteoarthritis
Keywords: knee osteoarthritis; bariatric surgery; weight loss; knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This project is a prospective observational study that will involve the participation of 25 volunteers that qualify for having knee osteoarthritis, are going to be having gastric bypass surgery and are willing to participate in this study which is designed to last up to two years. Potential candidates will be interviewed using a standard set of questions related to the study

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee is one of the five leading causes of disability among elderly men and women1. According to the American Academy of Orthopedic Surgeons, an estimated 19 million visits are made each year to physician's offices due to knee-related problems, while the total cost of OA was estimated at $60 billion in 2004.2

Obesity is a primary risk factor for the development of OA among several other features such as age, gender, trauma, infection, heredity, and high impact sports. In the United States, obesity has reached epidemic proportions and experiments have shown that individuals clinically defined as obese with a BMI > 30.0 kg/m2 are four times more likely to have knee OA than those with a BMI < 25.0 kg/m2(3).

The most common non-surgical treatment for knee OA has been the use of non-steroidal anti-inflammatory drugs (NSAIDs). NSAIDs work by inhibiting the cyclooxygenase (COX) enzymes involved in the production of pro-inflammatory molecules in the body. Although the use of these drugs has been shown to temporarily relieve pain and swelling associated with OA, there are several negative side-effects related to NSAID use including health concerns and cost.

If chronic NSAID use for knee pain can be reduced, that would be an exceptional public health benefit and would decrease cost and related hospital admissions and deaths.

This study investigates a non-surgical approach to the relief of pain associated with osteoarthritis in an attempt to offer a safer, less expensive alternative to other treatments.

In this study we will be examining the effect of weight loss through bariatric surgery on Knee pain in patients with clinical criteria indicative of osteoarthritis.

Our main objective is to determine if weight loss from bariatric surgery contributes to relief of knee pain and increased function in patients with osteoarthritis.

The study will be looking at obese patients with co-morbidity of knee osteoarthritis.

An interview will be administered and if appropriate, potential candidates will be asked a series of questions taken from the pain section of the Western Ontario McMaster Universities Index of Osteoarthritis (WOMAC). Patients with a WOMAC pain score ≥ 3 will then be asked to have a series of X-rays taken of their knees. Those individuals who display radiographic evidence of knee OA will be asked to participate in the study until the twenty five positions are filled. At their next pre-bariatric surgery visit, the study participants will have a basic knee exam performed by Kevin P. Black, M.D. in order to evaluate the structural integrity and alignment of the knee joint. The information gathered from the exam will serve as a baseline measure of knee function for the study. Prior to undergoing surgery, each of the 25 patients will be asked to complete a full version of the WOMAC survey and a separate, related survey the Knee and Osteoarthritis Outcome Score (KOOS). These surveys will be re-administered at 6, 12, and 24 months post-surgery in order to assess any changes in knee pain and function.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study, patients must be between the 18 and 70 years of age
* Completed a pre-surgery psychological evaluation, and have had intermittent knee pain for at least a year.
* The bariatric surgery requirement involves a bypass of the stomach.
* Standard of care guidelines for this surgery require that these patients' previous dieting attempts were without success
* Medical problems related to obesity, such as diabetes, sleep apnea, hypoventilation, and joint pain.
* Patients will have a WOMAC pain scale score > 3, according to the study by Miller, et al.
* Patients will have a standing AP, lateral and Merchant radiographic scan taken to confirm that they have OA.

Exclusion Criteria:

* Patients will be ineligible for the study if any of these criteria are not met.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be looking at obese patients with co-morbidity of knee osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Outcome measures will be determined with the WOMAC and KOOS surveys. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Rogers, M.D., Study Director — Penn State Milton S. Hershey Medical Center, Dept of Surgery
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] 1. Osteoarthritis of the Knee: State of the Condition. American Academy of Orthopedic Surgeons. 2004. http://www.aaos.org/Research/documents/oainfo_knee.asp.
- [Background] Buckwalter JA, Saltzman C, Brown T. The impact of osteoarthritis: implications for research. Clin Orthop Relat Res. 2004 Oct;(427 Suppl):S6-15. doi: 10.1097/01.blo.0000143938.30681.9d. PMID 15480076
- [Background] Miller GD, Nicklas BJ, Davis C, Loeser RF, Lenchik L, Messier SP. Intensive weight loss program improves physical function in older obese adults with knee osteoarthritis. Obesity (Silver Spring). 2006 Jul;14(7):1219-30. doi: 10.1038/oby.2006.139. PMID 16899803
- [Background] Banthin, J. S. and Zodet, M. Trends in the Use and Expenditures for COX-2 Inhibitors and Traditional Nonsteroidal Anti-inflammatory Drugs, 1997-2003. Statistical Brief #139. September 2006. Agency for Healthcare Research and Quality, Rockville, Md. http://www.meps.ahrq.gov/papers/st139/stat139.
- [Background] Blower AL, Brooks A, Fenn GC, Hill A, Pearce MY, Morant S, Bardhan KD. Emergency admissions for upper gastrointestinal disease and their relation to NSAID use. Aliment Pharmacol Ther. 1997 Apr;11(2):283-91. doi: 10.1046/j.1365-2036.1997.d01-604.x. PMID 9146764
- [Background] Graham GG, Graham RI, Day RO. Comparative analgesia, cardiovascular and renal effects of celecoxib, rofecoxib and acetaminophen (paracetamol). Curr Pharm Des. 2002;8(12):1063-75. doi: 10.2174/1381612023394917. PMID 11945151
- [Background] Aw TJ, Haas SJ, Liew D, Krum H. Meta-analysis of cyclooxygenase-2 inhibitors and their effects on blood pressure. Arch Intern Med. 2005 Mar 14;165(5):490-6. doi: 10.1001/archinte.165.5.IOI50013. Epub 2005 Feb 14. PMID 15710786